CLINICAL TRIAL: NCT03102697
Title: Optimization and Follow-up of the Consecutive Use of Two Intragastric Balloons (Heliosphere Bag®) in the Treatment of Obesity: A Prospective Clinical Study
Brief Title: Optimization and Follow-up of the Consecutive Use of Two Intragastric Balloons in the Treatment of Obesity
Status: Completed | Type: Observational
Sponsor: Kaiser Clinic and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: kaiserairballoonobesity
Record Dates: First submitted 2017-03-24; First posted 2017-04-06 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: Intragastric balloon; obesity; metabolic syndrome; bariatric surgery
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese individuals: Obese patients submitted to treatment using two consecutively air-filled IGB (Heliosphere® 600 cc and Heliosphere 720 cc) without any interval between the removal of the first and the placement of the second.
  Interventions: Device: Air-filled Intragastric balloon

INTERVENTIONS:
Device: Air-filled Intragastric balloon — Weight loss system that consists of an air balloon that occupies space in the stomach, thus reducing the gastric capacity and leaving less volume for food.
  Other Names: Heliosphere® 600 cc and Heliosphere 720 cc

SUMMARY:
This is a cohort study with the objective of describing during a 12-month follow-up, weight loss in obese patients submitted to treatment using two consecutively air-filled IGB (Heliosphere® 600 cc and Heliosphere 720 cc) without any interval between the removal of the first and the placement of the second.

DETAILED DESCRIPTION:
Intragastric balloon (IGB) implantation is a widely used technique to treat overweight subjects and those with mild obesity. The effectiveness of the air filled balloon (Heliosphere BAG®) in improving weight loss, reduction of BMI, percentage of body weight loss, percentage of excess weight loss and complications six months after placement is notable. Several methods are available for IGB placement and new techniques are being developed to reduce discomfort during and after the procedure. Thus, the use of an IGB as an effective method to avoid bariatric surgery is proposed. However, the precise protocol to balance complications and discomfort while maximizing weight loss is still to be established.

Our secondary objectives will be:

* Describe the weight loss, changes in the BMI and excess weight loss between the implantation of the first IGB until its removal;
* Describe changes in the components of the metabolic syndrome;
* Describe changes in blood pressure;
* Estimate the rate of early explant;
* Describe the conditions of surgery;
* Describe operative complications;
* To describe safety in the perioperative period, in the immediate postoperative period and in the late postoperative period

ELIGIBILITY:
Inclusion Criteria:

* Class I obesity (30-34.9 kg/m2), Class II obesity (35-39.5 kg/m2) or overweight (25-29.9 kg/m2).

Exclusion Criteria:

* Morbid obesity (BMI>40kg/m2), operative contraindications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese or overweight individuals eligible for gastric balloon placement and with no contraindications for the procedure will be recruited from the Mario Covas Hospital and the Kaiser Day Hospital.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Weight loss | 12 months
  Subtraction of the Final body mass index (BMI ) after 12 months of IGB placement minus the initial BMI

SECONDARY OUTCOMES:
Rate of early explant | 12 months
  Rate of patients in which the balloon was extracted early
Operative complications | Through endoscopy completion, an average of 2 hours
  Rate of complications during the placement of the balloon
Change in blood pressure | 12 months
  Arterial blood pressure will be measured before and after IGB using an digital sphygmomanometer
Changes Glycated hemoglobin (HbA1c) | 12 months
  Blood measurements of Glycated hemoglobin (HbAq1c) will be reported in International Federation of Clinical Chemistry and Laboratory Medicine Units
Physical activity | 12 months
  Physical activity will be self-reported on a weekly basis
Caloric intake | 12 months
  Caloric intake will be self-reported on a weekly basis
Excess weight loss | 12 months
  Measure that relates the preoperative weight, the postoperative weight and ideal weight
Posoperative complications | Through posToperative period completion, an average of 72 hours after the termination of surgery
  Rate of postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Grecco, MD, Study Chair — School of Medicine of ABC, Santo Andre/SP Brazil
Locations (1):
- School of Medice of ABC, Santo André, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided